CLINICAL TRIAL: NCT06829914
Title: Shockwave™ vs Surgical Endarterectomy for Calcified Severe Common Femoral Artery Stenosis: Comparison of Efficacy, Safety and Long-Term Outcomes
Acronym: Shockify
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 021-263
Record Dates: First submitted 2024-10-01; First posted 2025-02-17 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Common Femoral Artery Stenosis; Calcification; Heart
MeSH Terms: conditions — Calcinosis

STUDY DESIGN:
Intervention Model Description: Prospective, randomized pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Shockwave Catheter (Active Comparator): Shockwave™ Intravenous Lithotripsy (IVL)+ DCB (Drug Coated Balloon)
  Interventions: Device: Shockwave Catheter
- surgical endarterectomy (Active Comparator): Surgery should be performed with patch angioplasty, with or without profunda femoris endarterectomy.
  Interventions: Procedure: CFA Endarterectomy

INTERVENTIONS:
Device: Shockwave Catheter — Shockwave™ IVL + DCB procedure
  Arms: Shockwave Catheter
Procedure: CFA Endarterectomy — Standard CFA endarterectomy
  Arms: surgical endarterectomy

SUMMARY:
The investigators hypothesize that Shockwave with DCB is non-inferior to surgical endarterectomy for common femoral artery (CFA) stenosis with regard to primary efficacy and safety endpoints. The study will challenge the current guideline that recommends common femoral endarterectomy (CFE) as the primary treatment for symptomatic CFA stenosis.

DETAILED DESCRIPTION:
This is a pilot, prospective, randomized clinical trial. This trial compares patients with severe symptomatic moderate to severe calcified CFA stenosis undergoing traditional gold standard CFA endarterectomy to innovative technique of endovascular treatment using Shockwave™ Intra vascular Lithotripsy (IVL) using M5+ balloon with Drug coated balloon to achieve removal and debulking of plaque and achieve luminal gain. Patients who meet inclusion criteria will be informed and consented by a clinical coordinator if they wish to participate in the trial. If participants are candidates for surgery, they will then be randomized into one of two cohorts, receiving either Shockwave™ IVL + DCB (drug-coated balloon) procedure or a standard surgical endarterectomy. The study compares the 1-year efficacy and 6-month safety outcomes post-procedure for patients with severe, symptomatic CFA stenosis receiving Shockwave™ IVL with DCB versus surgical endarterectomy.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for inclusion in this study if he or she meets all of the following criteria (confirmed by core lab):

1. CFA atherosclerotic stenosis 60-100%
2. Moderate to severe calcification reported on imaging
3. Lifestyle-limiting intermittent claudication (IC) or chronic limb-threatening ischemia (CLTI) as described by Rutherford chronic limb ischemia (CLI) category 2-5
4. Failing conservative therapy
5. Operative candidate for CFE prior to enrollment
6. ≥18 years of age

Exclusion Criteria:

A patient will be ineligible for inclusion in this study if he or she meets any of the following criteria:

1. History of CFE or bypass in affected limb
2. Thrombosis of affected CFA
3. Aneurysm in the common femoral artery of target limb
4. Known target lesion restenosis (re-narrowing of the artery to ≥50% following the alleviation of a previous narrowing within 3 months)
5. Any preceding percutaneous cardiovascular intervention within 2 weeks
6. Inability to tolerate DAPT
7. Known coagulopathy or bleeding diathesis, thrombocytopenia with platelet count <100,000/µL
8. Uncontrolled diabetes (HbA1c ≥10.0%)
9. Non-ambulatory
10. Extensive tissue loss requiring amputation or salvageable only with complex foot reconstruction or non-traditional transmetatarsal amputations
11. MI within 6 weeks (defined as presumed ischemic symptoms (chest pain, ST-segment deviation and troponin higher than 2 times the upper limit of normal))
12. Stroke within 3 months (defined as sudden transient or irreversible focal neurological deficit resulting from a cerebrovascular cause)
13. Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2026-03-07 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Clinically driven target lesion revascularization (cdTLR (symptom-driven repeat revascularization of the index lesion)) | Procedure date through 1-year post-op
Restenosis to ≥ 50% of the target lesion on angiography or follow-up ultrasound | Procedure date through 1-year post-op
Freedom from perioperative death | Procedure date through 30 days post-op
Freedom from major adverse cardiovascular events (MACE (stroke, myocardial infarction (MI), cardiovascular death)) | Procedure date through 30 days post-op
Freedom from major adverse events | Procedure date through 6 months post-op
  1. Acute occlusion of the target lesion
  2. Flow-limiting dissection of the target lesion
  3. Symptomatic thrombus or embolus in treated limb requiring treatment
  4. Unplanned percutaneous/surgical revascularization or amputation above the ankle of the treated limb
  5. Access/surgical site complications
     1. Bleeding events (specify Bleeding Academic Research Consortium (BARC) type - see Appendix 18.2)
     2. Surgical site infection requiring medication or surgery, wound dehiscence, patch/arterial infection, lymphatic leak requiring surgery

SECONDARY OUTCOMES:
Mortality | Procedure date through 1-year post-op
Rutherford Chronic Limb Ischemia (CLI) Category | 30 days post-op, 3 months post-op, 6 months post-op, 1 year post-op
  https://www.ncbi.nlm.nih.gov/books/NBK553864/table/ch20.Tab2/#
  Stage 0 - Asymptomatic. Stage 1 - Mild claudication - Completes treadmill exercise; Ankle Pressure (AP) after exercise >50 mmHg but at least 20 mmHg lower than resting value.
  Stage 2 - Moderate claudication - Between categories 1 and 3. Stage 3 - Severe claudication - Cannot complete standard treadmill exercise and AP after exercise <50 mm Hg.
  Stage 4 - Ischemic rest pain - Resting AP <40 mm Hg, flat or barely pulsatile ankle or metatarsal pulse volume recording (PVR); Toe Pressure (TP) < 30 mm Hg.
  Stage 5 - Minor tissue loss-nonhealing ulcer, focal gangrene with diffuse pedal ischemia- Resting AP < 60 mm Hg, ankle or metatarsal PVR flat or barely pulsatile; TP < 40 mm Hg Stage 6 - Major tissue loss-extending above TM level, functional foot no longer salvageable - Same as category 5
Treatment satisfaction and quality of life (PAQ) | Pre-op, 30 days post-op, 6 months post-op, 1 year post-op
  Measured by the Peripheral Artery Questionnaire (PAQ), a 20-question questionnaire measuring peripheral vascular disease affect on quality of life. Questionnaires may be completed in-person or via phone call conducted by the study coordinator.
Intraoperative blood transfusion > 4 minutes | Intra-op
Procedural duration (minutes) | Intra-op
Length of stay (days) | Procedure date through 1 year post-op
Postoperative anemia requiring blood transfusion | Procedure date through 30 days post-op
Readmissions | 30 days post-op, 30 days post-discharge
Return to the operating room / angiography suite | 30 days post-op
Access/surgical site complications | 30 days post-op, 6 months post-op
  1. Superficial wound infection
  2. Deep wound infection
  3. Wound dehiscence
  4. Pseudoaneurysm identified on physical exam, imaging or angiography
  5. Hematoma identified on physical exam, imaging or angiography
Pneumonia (number of cases) | Procedure date through 30 days post-op
  Patients must meet criteria from both sections:
  Radiology: One definitive chest radiological exam (x-ray or CT) with at least one of the following:
  * New or progressive and persistent infiltrate
  * Consolidation or opacity
  Patients with underlying pulmonary or cardiac disease require two serial chest radiological exams (x-ray or CT) taken no less than 12 hours apart, but no more than 7 days apart.
  Signs/Symptoms/Laboratory: at least one of the following:
  * Fever (>38 C) with no other recognized cause
  * Leukopenia (<4000 WBC/mm3) or leukocytosis (≥12,000 WBC/mm3)
  * For adults ≥ 70 years old, altered mental status with no other recognized cause and at least one of the following:
    1. 5% Bronchoalveolar lavage (BAL)
    2. Positive growth in blood culture not related to another source of infection
    3. Positive growth in culture of pleural fluid
    4. Positive quantitative culture from minimally contaminated lower respiratory tract (LRT) specimen
Prolonged intubation | Procedure date through 30 days post-op
  Intubation greater than 48 hours postoperatively
Urinary tract infection | Procedure date through 30 days post-op
  Must meet one of the following TWO criteria within 30 days of the operation:
  * fever (>38C)
  * urgency
  * frequency
  * dysuria
  * suprapubic tenderness
  AND urine culture of >105 colonies/mL urine with no more than two species of organisms
  OR two of the following:
  * fever (>38C)
  * urgency
  * frequency
  * dysuria
  * suprapubic tenderness
  AND any of the following:
  * dipstick test positive for leukocyte esterase and/or nitrite
  * pyuria (>10WBCs/mL or >3 WBC/hpf of unspun urine)
  * organisms seen on Gram stain of unspun urine
  * two urine cultures with repeated isolation of the same uropathogen with >102 colonies/mL urine in non-voided specimen
  * urine culture with <105 colonies/mL urine of single uropathogen in patient being treated with appropriate antimicrobial therapy
  * physician's diagnosis
  * physician institutes appropriate antimicrobial therapy
Sepsis | Procedure date through 30 days post-op
  The disorder spectrum spans from relatively mild physiologic abnormalities to septic shock. The most significant level is reported using the following criteria: SIRS (Systemic Inflammatory Response Syndrome), clinically recognized by the presence of two or more of the following in the same time frame:
  Temp >38 degrees C or 90 bpm RR >20 breaths/min or PaCO2 12,000 cell/mm3, 10% immature (band) forms anion gap acidosis. Report if the patient has clinical signs and symptoms of SIRS listed above and meets either A or B:
  A. One of the following:
  * Positive blood culture
  * Clinical documentation of purulence or positive culture
  B. Suspected pre-operative infection or bowel infarction leading to the surgical procedure. Procedural findings must confirm this suspected diagnosis with one or more of the following:
  * Confirmed infarcted bowel requiring resection
  * Purulence in the operative site
  * Enteric contents in the operative site
  * Positive intra-operative cultures
Septic shock | Procedure date through 30 days post-op
  Report this variable if the patient has sepsis AND documented organ and/or circulatory dysfunction. Examples of organ dysfunction include: oliguria, acute alteration in mental status, acute respiratory distress. Examples of circulatory dysfunction include: hypotension, requirement of inotropic or vasopressor agents. The presence of pneumatosis along with the presence of SIRS is assigned.
Graft failure | Procedure date through 30 days post-op
  Mechanical failure of an extracardiac graft or prosthesis including myocutaneous flaps and skin grafts requiring return to the operating room, interventional radiology or a balloon angioplasty within 30 days of the operation.
Cardiac arrest | Procedure date through 30 days post-op
  The absence of cardiac rhythm or presence of chaotic cardiac rhythm, intraoperatively or postoperatively, which results in a cardiac arrest requiring the initiation of CPR, which includes chest compressions. Patients are included who are in a pulseless VT or Vfib in in which defibrillation is performed and PEA arrests requiring chest compressions. Patients with automated implantable cardioverter defibrillator (AICD) that fire but the patient has no loss of consciousness should be excluded.
Myocardial infarction | Procedure date through 30 days post-op
  Documentation of one or more of the following changes indicative of acute MI:
  * ST elevation >1mm in two or more contiguous leads
  * New left bundle branch block
  * New q-wave in two or more contiguous leads
  * New elevation in troponin greater than 3 times the upper level o f the reference range in the setting of suspected myocardial ischemia
Acute kidney injury | Procedure date through 30 days post-op
  In a patient who did not require dialysis preoperatively, worsening of renal dysfunction postoperatively requiring hemodialysis, peritoneal dialysis, hemofiltration, hemodiafiltration, or ultrafiltration
Dialysis | Procedure date through 30 days post-op
  Initiation of hemodialysis, peritoneal dialysis, hemofiltration, hemodiafiltration or ultrafiltration in a patient not previously on said therapy preoperatively
Deep vein thrombosis | Procedure date through 30 days post-op
  New diagnosis of blood clot or thrombus within the venous system (superficial or deep) which may be coupled with inflammation and requires treatment. Must be noted within 30 days after the principal operative procedure AND one of the following A or B below:
  A.New Diagnosis of a [new] venous thrombosis (superficial or deep), confirmed by a duplex, venogram, CT scan, or any other definitive imaging modality (including direct pathology examination such as autopsy) AND the patient must be treated with anticoagulation therapy and/or placement of a vena cava filter or clipping of the vena cava, or the record indicates that treatment was warranted but there was no additional appropriate treatment option available.
  B. As per (A) above, but the patient or decisionmaker has refused treatment. There must be documentation in the medical record of the [patient's] refusal of treatment.
Pulmonary embolism | Procedure date through 30 days post-op
  Lodging of a blood clot in the pulmonary artery with subsequent obstruction of blood supply to the lung parenchyma. The blood clots usually originate from the deep leg veins or pelvic venous system. Since there are not always preoperative studies proving that a clot or thrombus was not present preoperatively, the technical specification of the variable requires only a "new diagnosis"- in other words the clot or thrombus was not previously known. A pulmonary embolism must be noted within 30 days after the principal operative procedure AND the following criteria, A AND B below:
  A. New diagnosis of a new blood clot in a pulmonary artery
  AND
  B. The patient has a V-Q scan interpreted as high probability of pulmonary embolism or a positive CT exam, TEE, pulmonary arteriogram, CT angiogram, or any other definitive imaging modality (including direct pathology examination such as autopsy

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Sayfo, MD, Principal Investigator — Baylor Scott & White The Heart Hospital - Plano; John Kedora, MD, Principal Investigator — Baylor Scott & White The Heart Hospital - Plano
Locations (1):
- Baylor Scott & White The Heart Hospital - Plano, Plano, Texas, United States

REFERENCES:
- [Background] Kang JL, Patel VI, Conrad MF, Lamuraglia GM, Chung TK, Cambria RP. Common femoral artery occlusive disease: contemporary results following surgical endarterectomy. J Vasc Surg. 2008 Oct;48(4):872-7. doi: 10.1016/j.jvs.2008.05.025. Epub 2008 Jul 17. PMID 18639427
- [Background] Kuma S, Tanaka K, Ohmine T, Morisaki K, Kodama A, Guntani A, Ishida M, Okazaki J, Mii S. Clinical Outcome of Surgical Endarterectomy for Common Femoral Artery Occlusive Disease. Circ J. 2016;80(4):964-9. doi: 10.1253/circj.CJ-15-1177. Epub 2016 Feb 19. PMID 26902450
- [Background] Nguyen BN, Amdur RL, Abugideiri M, Rahbar R, Neville RF, Sidawy AN. Postoperative complications after common femoral endarterectomy. J Vasc Surg. 2015 Jun;61(6):1489-94.e1. doi: 10.1016/j.jvs.2015.01.024. Epub 2015 Feb 19. PMID 25702917
- [Background] Shammas NW, Abi Doumet A, Karia R, Khalafallah R. An Overview of the Treatment of Symptomatic Common Femoral Artery Lesions with a Focus on Endovascular Therapy. Vasc Health Risk Manag. 2020 Feb 20;16:67-73. doi: 10.2147/VHRM.S242291. eCollection 2020. PMID 32110032
- [Background] Bonvini RF, Rastan A, Sixt S, Noory E, Schwarz T, Frank U, Roffi M, Dorsaz PA, Schwarzwalder U, Burgelin K, Macharzina R, Zeller T. Endovascular treatment of common femoral artery disease: medium-term outcomes of 360 consecutive procedures. J Am Coll Cardiol. 2011 Aug 16;58(8):792-8. doi: 10.1016/j.jacc.2011.01.070. PMID 21835313
- [Background] Linni K, Ugurluoglu A, Hitzl W, Aspalter M, Holzenbein T. Bioabsorbable stent implantation vs. common femoral artery endarterectomy: early results of a randomized trial. J Endovasc Ther. 2014 Aug;21(4):493-502. doi: 10.1583/14-4699R.1. PMID 25101576
- [Background] Stavroulakis K, Schwindt A, Torsello G, Beropoulis E, Stachmann A, Hericks C, Bollenberg L, Bisdas T. Directional Atherectomy With Antirestenotic Therapy vs Drug-Coated Balloon Angioplasty Alone for Common Femoral Artery Atherosclerotic Disease. J Endovasc Ther. 2018 Feb;25(1):92-99. doi: 10.1177/1526602817748319. Epub 2017 Dec 18. PMID 29251204
- [Background] Garcia LA, Lyden SP. Atherectomy for infrainguinal peripheral artery disease. J Endovasc Ther. 2009 Apr;16(2 Suppl 2):II105-15. doi: 10.1583/08-2656.1. PMID 19624078
- [Background] Brodmann M, Werner M, Brinton TJ, Illindala U, Lansky A, Jaff MR, Holden A. Safety and Performance of Lithoplasty for Treatment of Calcified Peripheral Artery Lesions. J Am Coll Cardiol. 2017 Aug 15;70(7):908-910. doi: 10.1016/j.jacc.2017.06.022. No abstract available. PMID 28797363
- [Background] Brodmann M, Werner M, Holden A, Tepe G, Scheinert D, Schwindt A, Wolf F, Jaff M, Lansky A, Zeller T. Primary outcomes and mechanism of action of intravascular lithotripsy in calcified, femoropopliteal lesions: Results of Disrupt PAD II. Catheter Cardiovasc Interv. 2019 Feb 1;93(2):335-342. doi: 10.1002/ccd.27943. Epub 2018 Nov 25. PMID 30474206
- [Background] Adams G, Shammas N, Mangalmurti S, Bernardo NL, Miller WE, Soukas PA, Parikh SA, Armstrong EJ, Tepe G, Lansky A, Gray WA. Intravascular Lithotripsy for Treatment of Calcified Lower Extremity Arterial Stenosis: Initial Analysis of the Disrupt PAD III Study. J Endovasc Ther. 2020 Jun;27(3):473-480. doi: 10.1177/1526602820914598. Epub 2020 Apr 3. PMID 32242768
- [Background] Adams G, Soukas PA, Mehrle A, Bertolet B, Armstrong EJ. Intravascular Lithotripsy for Treatment of Calcified Infrapopliteal Lesions: Results from the Disrupt PAD III Observational Study. J Endovasc Ther. 2022 Feb;29(1):76-83. doi: 10.1177/15266028211032953. Epub 2021 Aug 12. PMID 34380334
- [Background] Baig M, Kwok M, Aldairi A, Imran HM, Khan MS, Moustafa A, Hyder ON, Saad M, Aronow HD, Soukas PA. Endovascular Intravascular Lithotripsy in the Treatment of Calcific Common Femoral Artery Disease: A Case Series With an 18-Month Follow-Up. Cardiovasc Revasc Med. 2022 Oct;43:80-84. doi: 10.1016/j.carrev.2022.05.003. Epub 2022 May 7. PMID 35595607
- [Background] Rutherford RB, Baker JD, Ernst C, Johnston KW, Porter JM, Ahn S, Jones DN. Recommended standards for reports dealing with lower extremity ischemia: revised version. J Vasc Surg. 1997 Sep;26(3):517-38. doi: 10.1016/s0741-5214(97)70045-4. PMID 9308598
- [Background] Tepe G, Brodmann M, Werner M, Bachinsky W, Holden A, Zeller T, Mangalmurti S, Nolte-Ernsting C, Bertolet B, Scheinert D, Gray WA; Disrupt PAD III Investigators. Intravascular Lithotripsy for Peripheral Artery Calcification: 30-Day Outcomes From the Randomized Disrupt PAD III Trial. JACC Cardiovasc Interv. 2021 Jun 28;14(12):1352-1361. doi: 10.1016/j.jcin.2021.04.010. PMID 34167675
- [Background] Varcoe RL, DeRubertis BG, Kolluri R, Krishnan P, Metzger DC, Bonaca MP, Shishehbor MH, Holden AH, Bajakian DR, Garcia LA, Kum SWC, Rundback J, Armstrong E, Lee JK, Khatib Y, Weinberg I, Garcia-Garcia HM, Ruster K, Teraphongphom NT, Zheng Y, Wang J, Jones-McMeans JM, Parikh SA; LIFE-BTK Investigators. Drug-Eluting Resorbable Scaffold versus Angioplasty for Infrapopliteal Artery Disease. N Engl J Med. 2024 Jan 4;390(1):9-19. doi: 10.1056/NEJMoa2305637. Epub 2023 Oct 25. PMID 37888915
- [Background] Spertus J, Jones P, Poler S, Rocha-Singh K. The peripheral artery questionnaire: a new disease-specific health status measure for patients with peripheral arterial disease. Am Heart J. 2004 Feb;147(2):301-8. doi: 10.1016/j.ahj.2003.08.001. PMID 14760329